CLINICAL TRIAL: NCT00724581
Title: Amiodarone Prophylaxis for Atrial Fibrillation in Patients Undergoing Surgery for Lung Cancer: A Controlled, Randomized, Double Blinded Trial
Brief Title: Amiodarone Prophylaxis for Atrial Fibrillation in Patients Undergoing Surgery for Lung Cancer
Acronym: PASCART
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Lars Riber Zebis, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2612-3681
Record Dates: First submitted 2008-07-25; First posted 2008-07-29 (Estimated); Last update posted 2008-07-29 (Estimated); Status verified 2008-07

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation, amiodarone
MeSH Terms: conditions — Atrial Fibrillation | interventions — Amiodarone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental)
  Interventions: Drug: Amiodarone

INTERVENTIONS:
Drug: Amiodarone — intravenous bolus of 300 mg oral treatment og 600 mg twice a day for five days

SUMMARY:
Patients undergoing lung resection due to pulmonary cancer can be compromised in their postoperative period due to atrial fibrillation.

A retrospective analysis performed at our institution indicates that 30 % of the population develope atrial fibrillation in the postoperative period.

Amiodarone is known to diminish the occurence of postoperative atrial fibrillation after heart surgery, why this drug is chosen as a prophylactic agent for the mentioned population.

Amiodarone is administrated twice a day for 5 days at a dose of 600 mg oral treatment after an initial loading bolus og 300 mg intravenously.

ELIGIBILITY:
Inclusion Criteria:

* Resection of the lung due to confirmed diagnosis of cancer pulmones.
* Elective operation (scheduled operation for at least one day)
* Ready to be randomized
* Patient must be at least 18 at time of operation

Exclusion Criteria:

* Former operation of the lung
* Former heart surgery
* Bradycardia below 40 beats/ min
* Hypotension with systolic blood pressure below 80 mmHg
* AV-blockage of any degree or sick sinus node
* QTc interval above 440 ms for men or above 460 ms for women
* Paroxysmal, persistent or permanent atrial fibrillation or flutter
* Former atrial fibrillation or flutter for more than a month.
* Pregnant or positive pregnancy test
* Breastfeeding
* ALAT of more than twice the normal over limit
* Treatment with monoamineoxidase inhibitors (MAOI)
* Allergy to one or more components in amiodarone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-08 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Free of atrial fibrillation | 31082009

SECONDARY OUTCOMES:
Cost-benefit analysis of amiodarone prophylactic | 31082009

CONTACTS AND LOCATIONS:
Overall Officials: Lars R Zebis, MD, Ph.D., Principal Investigator — Aarhus University Hospital Skejby
Locations (1):
- Aarhus University Hospital, Skejby, Aarhus, Denmark